CLINICAL TRIAL: NCT02816242
Title: Effect of Concept Mapping Teaching Method on Critical Thinking Skills of Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Ahvaz University of medical sciences (Unknown)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 94-5693
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Education
Keywords: Concept Map; critical thinking; medical student teaching

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): teaching anatomy by concept map
  Interventions: Other: concept map teaching
- placebo (Sham Comparator): teaching anatomy by traditional method
  Interventions: Other: traditional teaching

INTERVENTIONS:
Other: concept map teaching — teaching anatomy using concept map to improve critical thinking
  Arms: intervention
Other: traditional teaching — teaching anatomy using lecture
  Arms: placebo

SUMMARY:
effect of concept map in teaching critical thinking was done with randomized study

DETAILED DESCRIPTION:
This quasi-experimental study with two groups design and pre-posttest method was conducted at Ahvaz University of Medical Sciences in 2014. About 100 Medical Students of in their third semester were recruited for the study based on census. Participants were divided into two intervention and control groups by using random sampling and Random Number Table List. Students in the control group were lectured in Anatomy using traditional lecture method. Whereas, students in the experimental group were taught Anatomy using concept map teaching method. Student's critical thinking was evaluated by examining" Standard California Critical Thinking Skills Questionnaire"

ELIGIBILITY:
Inclusion Criteria:

* any student at 1st semester of medicine who accept participation in study

Exclusion Criteria:

* do not accepting to participate

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Standard California Critical Thinking Skills Questionnaire score | 4 months
  score which was got from questionnaire pre and post intervention

SECONDARY OUTCOMES:
student satisfaction | 4 months
  questionnaire for satisfaction
anatomy score | 4 months
  scores of anatomy in same exam at final

CONTACTS AND LOCATIONS:
Locations (1):
- Education Developmen Center, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No